CLINICAL TRIAL: NCT01316978
Title: A Single-Dose, Randomised, Crossover Bioequivalence Study to Compare the Rate and Extent of Absorption of a Test Formulation of Ibuprofen Fast Melt Orodispersible Tablet Versus Two Reference Formulations in Healthy Volunteers
Brief Title: A Study to Test Bioequivalence Between One Test Formulation of Ibuprofen and Two Reference Treatments
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: McNeil AB (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: IBUPAI1001
Record Dates: First submitted 2011-03-15; First posted 2011-03-16 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Experimental (Experimental): Experimental Ibuprofen
  Interventions: Drug: Ibuprofen
- Nurofen (Active Comparator): Nurofen Meltlets Orodispersible Tablet
  Interventions: Drug: Ibuprofen
- Motrin (Active Comparator): Junior Strength Motrin Chewable Tablet
  Interventions: Drug: Ibuprofen

INTERVENTIONS:
Drug: Ibuprofen — A single 2 x 100 mg dose of an experimental Ibuprofen Fast Melt Orodispersible Tablet administered orally, with a 7-day washout between visits
  Other Names: Not yet marketed
  Arms: Experimental
Drug: Ibuprofen — A single 200 mg Nurofen Meltlets Orodispersible Tablet administered orally, with a 7-day washout between visits
  Other Names: Nurofen Meltlets Orodispersible Tablet
  Arms: Nurofen
Drug: Ibuprofen — A single 2 x 100 mg dose of Junior Strength Motrin Chewable Tablet administered orally, with a 7-day washout between visits
  Other Names: Junior Strength Motrin Chewable Tablet
  Arms: Motrin

SUMMARY:
This study is designed to assess bioequivalence between one test and two reference formulations used for treatment of headaches and temporary relief of pain.

DETAILED DESCRIPTION:
The study is a single dose, randomized, three-way crossover study in 30 healthy subjects, with equal numbers of males and females (minimum of 13 of either gender). Drop-outs will not be replaced. The three doses of medication given in the study (a single dose in each of the three study periods) will each be separated by a washout period of at least 7 calendar days. In each study period, eighteen (18) blood samples for pharmacokinetic analysis will be taken over 12 hours. Blood samples will be centrifuged and concentrations of ibuprofen (R-enantiomer and S-enantiomer) in plasma will be measured using a validated chromatographic assay. Pharmacokinetic parameters will be calculated from plasma concentration data [R-enantiomer, S-enantiomer and total (sum of both enantiomers)]. The rate and extent of absorption of the formulations will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects (equal numbers of males and females)
* Volunteers aged of at least 18 years but not older than 55 years
* Subjects will have a Body Mass Index (BMI) greater than or equal to 18.5 and below 30 kg/m2; and a total body weight >50 kg
* Non- or ex-smokers; an ex-smoker being defined as someone who completely stopped smoking for at least 12 months before day 1 of this study.
* Clinical laboratory values within the laboratory's stated normal range; if not within this range, they must be without any clinical significance
* Have no clinically significant diseases captured in the medical history or evidence of clinically significant findings on physical examination and/or clinical laboratory evaluations (hematology, biochemistry, ECG and urinalysis)
* Has signed and dated the informed consent document, indicating that the subject has been informed of all pertinent aspects of the study
* Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures

Exclusion Criteria:

* Seated pulse rate below 45 bpm or higher than 90 bpm at screening
* Seated blood pressure below 90/60 mmHg or higher than 140/90 mmHg at screening
* Relationship to persons involved directly with the conduct of the study (i.e., principal investigator; sub-investigators; study coordinators; other study personnel; employees or contractors of the sponsor or Johnson & Johnson subsidiaries; and the families of each)
* Presence of any tongue piercings
* Presence of braces
* Females who are pregnant or are lactating
* Females of childbearing potential or males with a female partner of childbearing potential who refuse to use an acceptable contraceptive regimen throughout the entire duration of the study
* Females who are pregnant according to a positive serum pregnancy test
* Any medical history or condition, or use of any drug or medication, that the investigator determines could compromise subject safety or the evaluation of results.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2011-02; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration | During 12 hours post-dose
  Maximum Observed Plasma Concentration (Cmax), which is the maximum (peak) concentration (amount of drug) measurable in blood plasma after a dose is administered, measured in nanograms/milliliter (ng/mL)
Bioavailability [AUC(0-t)] | During 12 hours post-dose
  Bioavailability [AUC(0-t)] is a measure of how much of the drug reaches the person's bloodstream within a given period of time for the body to use. The extent of product bioavailability is estimated by the area under the blood concentration vs time curve. The Area Under the Curve (AUC) is calculated by plotting the drug's blood levels on a graph at different times during the set period. The area under this curve reflects the amount of drug exposure in the set time period, calculated as hour * nanograms (ng) per milliliter (mL).

SECONDARY OUTCOMES:
Bioavailability Extrapolated to Infinity [AUC (0-∞)] | 12 hours post-dose
  Bioavailability Extrapolated to Infinity [AUC (0-∞)] is a calculated measure of how much of the drug will ever reach the person's bloodstream for the body to use. AUC (0-∞) stands for the area under the plasma concentration versus time curve from time zero (pre-dose) to extrapolated infinite time (forever). It is obtained from calculating AUC (0-t) plus AUC (t-∞).
Time of Maximum Concentration | During 12 hours post-dose
  The time at which maximum concentration is reached (Tmax)
Terminal Elimination Rate Constant | During 12 hours post-dose
  The Terminal Elimination Rate Constant (Lamda z) is the time required to eliminate half the administered dose
Terminal Phase Plasma Half-Life | During 12 hours post-dose
  Terminal phase plasma half-life (t ½) is the time required to divide the plasma concentration by two after reaching pseudo-equilibrium, rather than the time required to eliminate half the administered dose.

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Kruse, PhD, Study Director — McNeil AB
Locations (1):
- Algorithme Pharma Inc., Mount Royal, Quebec, Canada